CLINICAL TRIAL: NCT06148454
Title: Implementation of Structured Positive Psychology Interventions to Improve Well-being and Resilience Amongst Anaesthesiologists in Hong Kong
Brief Title: Study of Positive Psychology and Effects on Well-being of Anaesthesiologists in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong College of Anaesthesiologists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PosPsychology1
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Burn Out; Stress, Psychological; Well-Being, Psychological; Self-Compassion; Depressive Symptoms; Anxiety Disorders and Symptoms
MeSH Terms: conditions — Burnout, Psychological; Stress, Psychological; Psychological Well-Being; Depression; Anxiety Disorders | interventions — Dilatation and Curettage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive Psychology A & B (Experimental): Module A and B
  Interventions: Behavioral: App-based Positive Psychology Intervention (A&B)
- Positive Psychology C & D (Experimental): Module C and D
  Interventions: Behavioral: App-based Positive Psychology Intervention (C&D)
- Control Group with no intervention (No Intervention)

INTERVENTIONS:
Behavioral: App-based Positive Psychology Intervention (A&B) — An app-based, evidence-based positive psychology intervention focusing on two modules: (A) Awareness & Positivity and (B) Meaning and Accomplishment
  Arms: Positive Psychology A & B
Behavioral: App-based Positive Psychology Intervention (C&D) — An app-based, evidence-based positive psychology intervention focusing on two modules: (C) Rapport & Conflict Management and (D) Compassion & Leadership
  Arms: Positive Psychology C & D

SUMMARY:
This clinical trial aims to evaluate whether positive psychology interventions via a hybrid approach will enhance well-being and resilience amongst anaesthesiologists in Hong Kong.

The main questions it aims to answer are:

* Is app-based positive psychology intervention effective in improving well-being of physicians?
* Is app-based positive psychology intervention feasible amongst busy healthcare professionals?

Participants will be randomized to one of the two groups:

* Four-week web-based interventions
* Control group

Researchers will compare the intervention and control groups to see if the participants' benefit from the positive psychology intervention compared with not receiving it.

ELIGIBILITY:
Inclusion Criteria:

* Fellows/members of The Hong Kong College of Anaesthesiologists

Exclusion Criteria:

* No exclusion criteria is applied

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported well-being | 4 weeks (Change from baseline to within 7 Days post-intervention)
  Overall well-being score of the Workplace PERMA-Profiler (Butler & Kern, 2016). This questionnaire consists of 23 items on a 10-point Likert scale from 0 = not at all to 10 = completely. The scale measures five pillars of well-being: positive emotion (P), engagement (E), relationship (R), meaning (M), and accomplishment (A), along with filler questions measuring negative emotion (N) and health (H). A overall well-being score is calculated to represent the person's well-being.
Self-reported burnout | 4 weeks (Change from baseline to within 7 Days post-intervention)
  Overall burnout score of Copenhagen Burnout Inventory (CBI) (Kristensen, Borritz, Villadsen, & Christensen, 2005). This questionnaire consists of 19 items on a 5-point Likert scale from 1 = 0% (Never or almost never/To a very low degree) to 5 = 100% (Always/To a very high degree). The scale measures three domain of burnout: personal burnout, work-related burnout, and client-related burnout. A overall burnout score is calculated to represent the person's level of burnout.
Self-reported psychological stress | 4 weeks (Change from baseline to within 7 Days post-intervention)
  Total stress score of Perceived Stress Scale (PSS-10) (Cohen et al., 1983). This questionnaire consists of 10 items on a 5-point Likert scale from 0 = Never to 4 = Very Often. The scale has two subscales: perceived helplessness and lack of self-efficacy. A total stress score is calculated to represent the person's level of psychological stress.
Self-reported anxiety symptom | 4 weeks (Change from baseline to within 7 Days post-intervention)
  Total score of General Anxiety Disorder-7 (GAD-7) (Spitzer, Kroenke, Williams, & Löwe, 2006). This questionnaire consists of 7 items on a 4-point Likert scale from 0 = Not at all to 3 = Nearly every day. A total stress score is calculated to represent the person's anxiety symptom severity.
Self-reported depression symptom | 4 weeks (Change from baseline to within 7 Days post-intervention)
  Total score of Patient Health Questionnaire-9 (PHQ-9) (Kroenke, Spitzer, & Williams, 2001). This questionnaire consists of 9 items on a 4-point Likert scale from 0 = Not at all to 3 = Nearly every day. A total stress score is calculated to represent the person's depression symptom severity.

SECONDARY OUTCOMES:
Self-reported self-compassion | 4 weeks (Change from baseline to within 7 Days post-intervention)
  Self-Compassion Scale - Short Form (SCS-SF) (Raes, Pommier, Neff, & Van Gucht, 2011). This questionnaire consists of 12 items on a 5-point Likert scale from 1 = Strongly disagree to 5 = Strongly agree. The scale has six subscales: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. A total self-compassion score is calculated to represent the person's level of self-compassion.
Self-reported work gratitude | 4 weeks (Change from baseline to within 7 Days post-intervention)
  Overall gratitude at work score of Work Gratitude Scale (Youssef-Morgan, van Zyl, & Ahrens, 2022). This questionnaire consists of 10 items on a 7-point Likert scale from 1 = Almost never to 7 = Almost always. The scale measures three components gratitude at work: grateful appraisals, gratitude toward others, and intentional attiude of gratitude. An overall gratitude at work score is calculated to represent the person's gratitude in one's work setting.
Self-reported work meaning | 4 weeks (Change from baseline to within 7 Days post-intervention)
  Meaningful Work score of the Work and Meaning Inventory (Steger, Dik, & Duffy, 2012). This questionnaire consists of 10 items on a 5-point Likert scale from 1 = Absolutely untrue to 5 = Absolutely true. The scale has six subscales: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. A overall Meaningful work score is calculated to represent the depth to which the person experience their work as meaningful, as something they are personally invested in, and which is a source of flourishing in one's life.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Kam Ming Chan, Principal Investigator — The Hong Kong College of Anaesthesiologists
Locations (1):
- The Hong Kong College of Anaesthesiologists, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No